CLINICAL TRIAL: NCT04796350
Title: Randomized Controlled Study of a Local Osteo-Enhancement Procedure (LOEP) to Prevent Secondary Hip Fractures in Osteoporotic Women Undergoing Treatment of Index Hip Fractures
Brief Title: RESTORE - Study of AGN1 LOEP to Prevent Secondary Hip Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AgNovos Healthcare, LLC (Industry)
Collaborators: Avania (Industry); CMIC Co, Ltd. Japan (Industry); BioClinica, Inc. (Industry); Emergent Clinical Consulting, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AGN-CIP-100 / AGN-CIP-100-CA
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Fragility Fracture; Hip Fractures; Osteoporosis
Keywords: Osteoporosis; Hip Fracture; Fragility Fracture; LOEP; RESTORE; Local osteo-enhancement procedure
MeSH Terms: conditions — Hip Fractures; Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated group (Experimental): Subject receives standard of care to repair the index hip fracture and AGN1 LOEP treatment on the target unfractured contralateral hip
  Interventions: Device: AGN1 LOEP treatment
- Control group (No Intervention): Subject receives standard of care to repair the index hip fracture and no AGN1 LOEP treatment on the target unfractured contralateral hip

INTERVENTIONS:
Device: AGN1 LOEP treatment — the implantation site is injected with the AGN1 implant material
  Arms: Treated group

SUMMARY:
A randomized controlled trial to evaluate AGN1 to prevent secondary hip fractures in osteoporotic women undergoing treatment of index hip fractures. Up to 2400 subjects will be randomized between a treatment group and a control group. Subjects will be followed for a minimum of 5 years after undergoing hip fracture repair surgery.

DETAILED DESCRIPTION:
This is an event driven, randomized, controlled, prospective, single blinded (non-blinded in Canada), multi-national study.

This study is designed to demonstrate that the AGN1 LOEP treatment can reduce the incidence of secondary hip fractures in subjects presenting with an index hip fracture and undergoing hip fracture repair surgery. Subjects presenting with an index fragility hip fracture who will undergo hip fracture repair will be enrolled. Subjects will be randomized 1:1 into the following two study groups:

1. Treated Group - receives standard of care to repair the index hip fracture and AGN1 LOEP treatment on the target unfractured contralateral hip
2. Control Group - receives standard of care to repair the index hip fracture and no AGN1 LOEP treatment on the target unfractured contralateral hip

AGN1 LOEP is an elective procedure that will be performed immediately following hip fracture repair.

Subjects will be followed through scheduled visits conducted at 6 weeks, 6 months, and every 6 months thereafter for a minimum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a postmenopausal female at least 1-year post menses and at least 65 years of age.
2. Subject presents with a low-energy index fragility hip fracture in one hip and will undergo surgical repair of the fractured hip.
3. Subject has at least one of the following additional risk factors for a secondary hip fracture (as determined by subject or legally authorized representative (LAR) interview or medical record review):

   * Documented falls assessment indicating subject is at moderate or high risk of falls
   * Falls history (2 or more falls in the previous 12 months)
   * History of vertigo, dizziness, or postural hypotension
   * Documented T-score < -2.5 at the hip
   * Taking more than 3 daily prescription medications
   * Visual impairment as confirmed by one of the following:

     * Subject reports difficulty seeing
     * Lack of depth perception or vision loss in one eye
     * Macular degeneration
     * Cataracts
   * Prior non-hip fragility fracture
   * Cognitive frailty as assessed by SPMSQ (mild or moderate cognitive impairment) or delirium
   * Parkinson's disease stage 3 or 4
   * 10-year hip fracture probability >15% using the FRAX® Fracture Risk Assessment Tool of the clinical site country
4. Subject is expected to be ambulatory after the hip fracture repair procedure.
5. Informed consent is provided by the subject or the subject's LAR.
6. The subject's willingness, ability, and commitment to participate in screening, treatment, and all follow-up evaluations for the full duration of the study has been documented.

Exclusion Criteria:

1. Subject hospital admission is > 24 hours from the time of the index hip fracture.
2. Subject was dependent on the use of a wheelchair or was bedridden prior to the index hip fracture.
3. Subject is currently enrolled in another clinical study.
4. Subject has a history of hip surgery or previous hip fracture on the target unfractured hip contralateral to the index hip fracture.
5. Subject has one or more new fractures in addition to the index hip fracture at admission that, in the opinion of the investigator, would further compromise patient mobility, rehabilitation, and/or recovery or subject has three or more new fractures in addition to the index hip fracture.
6. Subject has an infection at the LOEP intended treatment site or has non-intact skin or acute traumatic injuries with open wounds close to the area of intended LOEP treatment.
7. Subject has a progressive increase in undiagnosed pain in the target hip contralateral to the index fractured hip over the previous 3 months that in the opinion of the Investigator may suggest underlying bone or joint pathology on the unfractured side.
8. Subject has radiological evidence of gross bony or joint pathology of the hip, including signs predictive of atypical femoral fractures (e.g. cortical beaking), or has been diagnosed and/or treated for atypical femoral fractures.
9. Subject is at ASA Class IV, V, or VI.
10. Subject has a history of metabolic bone disease other than osteoporosis (e.g., Paget's disease, renal osteodystrophy, or osteomalacia).
11. Subject has a history of Pott's disease.
12. Subject has a history of any invasive malignancy (except nonmelanoma skin cancer), unless treated with curative intent and with no clinical signs or symptoms of the malignancy for 5 years.
13. Subject has chronic cardiac insufficiency or severe cardiovascular disease as assessed by a subject or LAR interview to be NYHA Class III or IV or has an implanted pacemaker.
14. Subject has a history of cardiovascular events (e.g. stroke, transient ischemic attack, myocardial infarction, unstable angina, pulmonary embolus, deep vein thrombosis, ventricular tachycardia, or atrial fibrillation) in the last 3 months.
15. Subject is on oral or parenteral immuno-suppressive drugs.
16. Subject has uncontrolled diabetes mellitus.
17. Subject has Hb ≤ 9 g/dL at admission.
18. Subject has severe renal insufficiency defined as an estimated glomerular filtration rate (eGFR) ≤ 30 mL/min.
19. Subject has a diagnosed and ongoing calcium metabolism disorder.
20. Subject has a Parker Mobility Score ≤ 5.
21. Subject has severe cognitive impairment as assessed by SPMSQ.
22. Subject has known allergies to calcium-based bone void fillers.
23. In the judgement of the Investigator, the subject is not a good study candidate (e.g., inability to maintain follow-up schedule, comorbidity or poor general physical/mental health, or drug or alcohol abuse issues).
24. Subject fails pre-operative or intraoperative eligibility criteria as specified in section 7.4.2. of the clinical investigation plan.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2021-04-24 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of secondary fragility hip fractures | Interim Analysis, approximately 30 Months
  Comparison of incidence of secondary fragility hip fractures in the target hip among the Treated Group vs. Control Group.
Cumulative Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Interim Analysis, approximately 30 Months
  Comparison of incidence of AEs and SAEs among the Treated Group vs. Control Group.

SECONDARY OUTCOMES:
Areal bone mineral density (aBMD) | 12 months and 24 months
  Total hip areal bone mineral density in target hips of the Treated Group compared to the Control Group
Trabecular Bone Score (TBS) | 12 months and 24 months
  Continuous densitometry measure of the target hip bone of the Treated Group compared to the Control Group

CONTACTS AND LOCATIONS:
Locations (54):
- Innsbruck Hospital, Innsbruck, Austria
- Health Sciences Centre - Eastern Health, St. John's, Newfoundland and Labrador, Canada
- Aarhus University Hospital, Aarhus, Denmark
- France (3):
  - CHU Grenoble-Alpes, Grenoble
  - CHU Lyon, Lyon
  - CHU Toulouse, Toulouse
- Germany (9):
  - University Hospital of Duesseldorf, Düsseldorf
  - Justus Liebig Universitat Gießen, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Klinikum der Universität München, München
  - University Hospital of Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - BG Klinik Tuebingen, Tübingen
  - Helios Wuppertal, Wuppertal
- Italy (5):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - ASST Gaetano Pini CTO, Milan
  - University Hospital San Raffaele Milano, Milan
  - Policlinico Tor Vergata, Rome
  - CTO Torino, Torino
- Japan (16):
  - Akita City Hospital, Akita, Akita
  - Southern Tohoku General Hospital, Kōriyama, Fukushima
  - Hyogo Prefectural Nishinomiya Hospital, Nishinomiya, Hyōgo
  - Kagawa Rosai Hospital, Marugame, Kagawa-ken
  - Kanto Rosai Hospital, Kawasaki, Kanagawa
  - Shin-yurigaoka General Hospital, Kawasaki-Shi, Kanagawa
  - Chikamori Hospital, Kochi, Kochi
  - Okayama Medical Center, Okayama, Okayama-ken
  - Jutendo University Shizuoka Hospital, Izunokuni, Shizuoka
  - The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - St. Mary's Hospital, Fukuoka
  - Iwata City Hospital, Iwata
  - Shin-Yurigaoka General Hospital, Kawasaki-shi
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Saga-Ken Medical Centre Koseikan, Saga
  - Japanese Red Cross Shizuoka Hospital, Shizuoka
- Netherlands (4):
  - Deventer Hospital, Deventer
  - Saint Anna Ziekenhuis, Geldrop
  - Maastricht UMC, Maastricht
  - Isala Hospital, Zwolle
- Spain (10):
  - Vall d'Hebron University Hospital, Barcelona, Barcelona
  - Valladolid University Clinic Hospital, Valladolid, Valladolid
  - Clinic de Barcelona, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Galdakao-Usansolo Hospital, Galdakao
  - Hospital Neuro-Traumatológico de Jaén, Jaén
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - PARC Tauli, Sabadell
  - Mutua de Terrassa University Hospital, Terrassa
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Nottingham University Hospitals, Queen's Medical Center, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Japan Registry of Clinical Trials — https://jrct.niph.go.jp/en-latest-detail/jRCT2022210008